CLINICAL TRIAL: NCT05589987
Title: Community's Participation of Children With Spinal Muscular Atrophy Using Power Mobility
Brief Title: Spinal Muscular Atrophy on Wheels, Using Power Mobility
Acronym: SMAPmob
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Castilla-La Mancha (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Rpalomo03
Record Dates: First submitted 2022-10-10; First posted 2022-10-21 (Actual); Last update posted 2022-10-21 (Actual); Status verified 2022-10

CONDITIONS: Spinal Muscular Atrophy
Keywords: home; family; natural environment; participation
MeSH Terms: conditions — Muscular Atrophy, Spinal

STUDY DESIGN:
Intervention Model Description: 2 groups: experimental and control groups.
Who Masked: Outcomes Assessor
Masking Description: the masking will be of the evaluator. The assessments will be passed by a study evaluator and scored by an evaluator external to the study to ensure blinding of the groups.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Power mobility (Experimental): The study will take place in the child's natural environment for 12 weeks.
  Interventions: Device: power mobility
- Non-power mobility (No Intervention): Children will perform their typical daily routine without any modification. After the study they will be invited to participate in the experimental group if positive benefits are obtained.

INTERVENTIONS:
Device: power mobility — Sessions of adjustment, adaptation and choice of the device for training will be carried out. Once the cars are fully adapted and conditioned to the environment and needs of the family and the child, the intervention will begin.
  The study will take place in the child's natural environment for 12 weeks. Three 40-minute sessions per week will be held, each session includes: 1) configuration of the environment (families will be instructed by the therapists to adapt the environment to the child's situation and their conditions for driving the car): 5 min ; 2) natural play as a warm-up activity: 5 min; and 3) mobility and social training with cars: 30 min. The 30-minute driving session will involve participants learning cause and effect concepts by driving the toy car (press the button to move and release to stop). The therapist and caregivers will use verbal cues to encourage children to drive and explore the environment. All sessions will be video and audio recorded.
  Arms: Power mobility

SUMMARY:
The group of children diagnosed with Spinal Muscular Atrophy (SMA) has serious restrictions on participation. SMA is a neuromuscular disease that leads to neuromusculoskeletal disorders that limit functional activities, sometimes making it impossible to sit down autonomously and to walk.

Scientific evidence has highlighted the importance of implementing physiotherapy interventions in pediatrics that facilitate the integration and participation of children with reduced mobility in their natural environment through the use of different assisted mobility devices that allow the child to acquire a degree of independence and motivation according to their potential and needs.

For some time, with the aim of offering independent movement opportunities for children with severe motor impairment, adapted electric cars have been used, as they are simple to use and easy for the child and family to incorporate into daily tasks within natural environments. These low-cost motorized devices can generate a very positive impact on the participation of children diagnosed with SMA type I from an early age, after training the family and/or the child himself, guaranteeing the maximum possible safety, comfort, motivation and autonomy.

Due to the above, there is a need to carry out the research project defined below, to generate opportunities for the inclusion of children diagnosed with SMA type I through the use of low-cost electric cars that encourage their participation, motivation and quality of life.

DETAILED DESCRIPTION:
OBJECTIVES

1. To know the acceptability of an intervention with motorized mobility through electric cars for young children diagnosed with SMA type I.
2. To check the effectiveness of the motorized mobility intervention with electric cars with respect to: (a) mobility and (b) participation of young children with SMA type I with respect to the control group of children who do not use such devices.
3. To identify the barriers and facilitators of the child's participation in their natural environment of a motorized mobility intervention with electric cars in young children with SMA type I.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of SMA type I
* Ages between 10 months to 5 years.
* No previous experience with motorized mobility.

Exclusion Criteria:

* severe visual problems
* Associated disorders that do not correspond to the diagnosis of SMA type I.
* Families who do not agree to have training in the use of the electric car and continuous monitoring by the corresponding researcher.

Ages: 10 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-11-30 (Estimated); Study Completion 2024-02-01 (Estimated)

PRIMARY OUTCOMES:
QUEST (Version 2.0) Quebec User Evaluation of Satisfaction with assistive Technology | baseline and Change from basaline at week 12
  the scale includes 12 items rated on a 5-point satisfaction scale. approximately 10-15 minutes are require to complete the evaluation.
YC-PEM (Young Children's Participation & Environment Measure) | baseline, Change from basaline at week 12 and Change from basaline at week 16
  to be used for children from zero to five years, explores the frequency of participation in activities. Parents will report their child's participation across home, community and childcare
Pediatric Evaluation of Disability Inventory-Computer Adaptive-test (PEDI-CAT) | baseline, Change from basaline at week 12 and Change from basaline at week 16
  It is answered by the children's caregiver and has an item bank divided into two domains:
  (1) mobility, which includes 75 items ranging from basic motor skills (e.g., sitting without support) to more difficult motor skills (e.g., running or climbing a step ladder). Additionally, this domain includes the use of walking devices; (2) cognitive/social, which includes 60 items related to interaction (e.g., follows the gaze of another person), communication (e.g., uses gestures to ask for something), everyday cognition (e.g., recognizes his/her name), and self-management (e.g., when upset response without hitting). In these domains, the four-point scores (unable, hard, a little hard, easy) are based on different levels of difficulty. The overall score is transformed in a normative score (based on age) and a continuous score that will be used in the analyses.
Photovoice | baseline,Change from basaline at week 12
  to record and present everyday realities using photography; promote dialogue and critical reflection of reality and know the strengths and weaknesses of the target audience; and reach decision makers

SECONDARY OUTCOMES:
Goal Attainment Scaling (GAS) | baseline, Change from basaline at week 12
  GAS is an objective method of quantifying goal attainment. Goals are scored on a Likert-type scale from -2 (representing no positive change at all from baseline/ regression), -1 (a little less change than expected), 0 (attainment of goal at the expected level), +1 (a little more change than expected), to +2 (attainment of goal at much more than the expected level)
Switch Activation | at the end of week 4, 8, and week 12
  Switch activation is defined as when the switch is pressed to activate the modified ride-on car and make it "go", thereby moving in space from one place to another
Daily driving journal | baseline, week 12 and week 16
  Parents will record the date, duration (minutes) location, and activities during each driving session in a daily driving journal.

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Rocío Castilla-La Palomo-Carrión, Toledo, Castilla-La Mancha/Toledo
  - University of Castilla-La Mancha, Toledo

IPD SHARING:
Plan to Share IPD: Undecided
we will share the data when researchers ask us about that

REFERENCES:
- [Result] Arnold WD, Kassar D, Kissel JT. Spinal muscular atrophy: diagnosis and management in a new therapeutic era. Muscle Nerve. 2015 Feb;51(2):157-67. doi: 10.1002/mus.24497. Epub 2014 Dec 16. PMID 25346245
- [Result] Livingstone R, Field D. Systematic review of power mobility outcomes for infants, children and adolescents with mobility limitations. Clin Rehabil. 2014 Oct;28(10):954-64. doi: 10.1177/0269215514531262. Epub 2014 Apr 24. PMID 24764156
- [Result] Feldner HA, Logan SW, Galloway JC. Why the time is right for a radical paradigm shift in early powered mobility: the role of powered mobility technology devices, policy and stakeholders. Disabil Rehabil Assist Technol. 2016 Feb;11(2):89-102. doi: 10.3109/17483107.2015.1079651. Epub 2015 Sep 4. PMID 26340446
- [Result] Ostensjo S, Carlberg EB, Vollestad NK. The use and impact of assistive devices and other environmental modifications on everyday activities and care in young children with cerebral palsy. Disabil Rehabil. 2005 Jul 22;27(14):849-61. doi: 10.1080/09638280400018619. PMID 16096237
- [Result] Demers L, Weiss-Lambrou R, Ska B. Item analysis of the Quebec User Evaluation of Satisfaction with Assistive Technology (QUEST). Assist Technol. 2000;12(2):96-105. doi: 10.1080/10400435.2000.10132015. PMID 11508406
- [Result] St John BM, Hladik E, Romaniak HC, Ausderau KK. Understanding health disparities for individuals with intellectual disability using photovoice. Scand J Occup Ther. 2018 Sep;25(5):371-381. doi: 10.1080/11038128.2018.1502349. Epub 2018 Oct 3. PMID 30280952
- [Result] Krasny-Pacini A, Hiebel J, Pauly F, Godon S, Chevignard M. Goal attainment scaling in rehabilitation: a literature-based update. Ann Phys Rehabil Med. 2013 Apr;56(3):212-30. doi: 10.1016/j.rehab.2013.02.002. Epub 2013 Feb 28. PMID 23562111
- [Result] Di Marino E, Tremblay S, Khetani M, Anaby D. The effect of child, family and environmental factors on the participation of young children with disabilities. Disabil Health J. 2018 Jan;11(1):36-42. doi: 10.1016/j.dhjo.2017.05.005. Epub 2017 Jun 1. PMID 28624289
- [Result] Haley SM, Coster WJ, Dumas HM, Fragala-Pinkham MA, Kramer J, Ni P, Tian F, Kao YC, Moed R, Ludlow LH. Accuracy and precision of the Pediatric Evaluation of Disability Inventory computer-adaptive tests (PEDI-CAT). Dev Med Child Neurol. 2011 Dec;53(12):1100-6. doi: 10.1111/j.1469-8749.2011.04107.x. Epub 2011 Nov 11. PMID 22077695